CLINICAL TRIAL: NCT03982238
Title: Effects of Continuous Subcutaneous Insulin Infusion and Oral Hypoglycemic Drugs on Testosterone Levels in Type 2 Diabetes Patients
Brief Title: Effects of Hypoglycemic Drugs on Testosterone Levels in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Majianhua (Other)
Responsible Party: Sponsor-Investigator, Majianhua, Director, Head of Endocrinology department, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20190530-12
Record Dates: First submitted 2019-06-09; First posted 2019-06-11 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Metformin; dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): continuous subcutaneous insulin infusion therapy
  Interventions: Drug: Insulin
- Metformin (Experimental): metformin therapy
  Interventions: Drug: Metformin
- Dapagliflozin (Experimental): Dapagliflozin
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Insulin — Continuous subcutaneous insulin infusion therapy for 1 month
  Arms: Control group
Drug: Metformin — Continuous subcutaneous insulin infusion plus metformin (at least1000mg/day) for 1 month
  Arms: Metformin
Drug: Dapagliflozin — Continuous subcutaneous insulin infusion plus metformin (10mg/day) for 1 month
  Arms: Dapagliflozin

SUMMARY:
The study will assess the total testosterone and sex hormone-binding globulin levels in men with type 2 diabetes before and after continuous subcutaneous insulin infusion and hypoglycemic drugs treatment.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes, aged 18-60 years old, meeting WHO1999 diagnostic criteria, have not used any hypoglycemic drugs.
* HbA1c > 9%.
* subjects are able and willing to eat and exercise regularly.

Exclusion Criteria:

* patients with insulin allergy.
* impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal.● drug abuse and alcohol dependence in the past 5 years.
* systemic hormone therapy was used in the last three months.
* patients with poor compliance and irregular diet and exercise.
* patients with infection and stress within 4 weeks.
* any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
total testosterone levels | 1 month
  changes of total testosterone levels

SECONDARY OUTCOMES:
bioavailable testosterone | 1 month
  changes of bioavailable testosterone
free testosterone | 1 month
  changes of free testosterone

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hu Y, Ding B, Shen Y, Yan RN, Li FF, Sun R, Jing T, Lee KO, Ma JH. Rapid Changes in Serum Testosterone in Men With Newly Diagnosed Type 2 Diabetes With Intensive Insulin and Metformin. Diabetes Care. 2021 Apr;44(4):1059-1061. doi: 10.2337/dc20-1558. Epub 2021 Feb 3. PMID 33536253